CLINICAL TRIAL: NCT06075511
Title: Prospective Study to Assess Fitness in Patients with Renal Failure Undergoing Sleeve Gastrectomy - PROFIT
Brief Title: A Study of Sleeve Gastrectomy Risks and Benefits
Status: Withdrawn | Type: Observational
Why Stopped: Funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aleksandra Kukla, Principal Investigator, Mayo Clinic
Other Study IDs: 23-002715
Record Dates: First submitted 2023-09-28; First posted 2023-10-10 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Renal Failure
Keywords: Sleeve Gastrectomy
MeSH Terms: conditions — Renal Insufficiency | interventions — Fitness Trackers; Blood Pressure Monitors; Blood Pressure Monitoring, Ambulatory; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples will be collected at baseline and 12 months for future studies s)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Renal Failure Sleeve Gastrectomy: Subjects that have renal failure and are undergoing a sleeve gastrectomy per standard clinical care will perform a 6-minute walk distance (6MWD) evaluation, activity monitoring, continuous glucose monitor (CGM), blood pressure monitoring, complete mixed meal test, and composition body scan to gather additional information for researchers.
  Interventions: Diagnostic Test: 6 minutes walk distance; Behavioral: Activity Monitor; Behavioral: Continuous Glucose Monitor; Behavioral: Blood Pressure Monitoring; Diagnostic Test: Blood Pressure Monitoring; Diagnostic Test: Body Composition Scan; Diagnostic Test: Mixed meal testing; Diagnostic Test: Quality of Life

INTERVENTIONS:
Diagnostic Test: 6 minutes walk distance — Subjects walk as far as possible for 6 minutes at a self-selected pace, and the total distance walked will be recorded
  Other Names: 6MWD
Behavioral: Activity Monitor — Subjects will wear an Actigraph on their wrist like a watch for up to 10 days at home to monitor activity.
Behavioral: Continuous Glucose Monitor — Subjects will collect glucose values in the fluid under their skin for up to 10 days at home.
  Other Names: CGM
Behavioral: Blood Pressure Monitoring — Subjects will monitor their blood pressure at home for 10 consecutive days 3 times a day
Diagnostic Test: Blood Pressure Monitoring — 24-hour ambulatory blood pressure monitoring
Diagnostic Test: Body Composition Scan — Measure of body fat percentage, skeletal muscle mass, body water, and visceral fat.
  Other Names: DEXA Scan
Diagnostic Test: Mixed meal testing — Subjects will consume 6 ml/kg body weight of Boost, up to maximum of 360 ml, within 5 min
Diagnostic Test: Quality of Life — Subject will complete Quality of Life Questionnaire
  Other Names: PROMIS Questionnaire

SUMMARY:
This research study is being conducted to collect information to improve the outcomes of patients who have renal failure and are scheduled to have a sleeve gastrectomy.

DETAILED DESCRIPTION:
We will collect information on changes in physical performance, activity, blood pressure and glucose metabolism, body composition, and the quality of life prior to and three months after sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant candidates with obesity.
* Accepted for sleeve gastrectomy (SG).
* Accepted for kidney transplantation if criteria are met after SG.

Exclusion Criteria:

* Not undergoing sleeve gastrectomy.
* Unable to connect through telehealth technology.
* History of medical non-adherence that can affect adherence to the protocol.
* Any other medical condition that in the opinion of the Principal Investigators warrants exclusion for safety reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified through the clinical setting that are diagnosed renal failure and scheduled for sleeve gastrectomy per standard of clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walk distance (6MWD) | Baseline, 12 weeks
  Total distance walked at a self-selected pace reported in meters

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) score | Baseline, 12 weeks
  Measure of physical performance through balance, strength, and gait measurements. Total score ranges for 0 = worst performance and 12 = best performance.
Change in total step count | Baseline, 12 weeks
  Total number of steps taken as measured by ActiGraph
Change in quality of life | Baseline, 12 weeks
  Assessed by the PROMIS 29 questionnaire to assess seven health domains (physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference) on an individual scoring scale of 1-5 where 1= not all all and 5= very much.
Change in glucose metrics | Baseline, 12 weeks
  Assessed by continuous glucose metabolism.
change in insulin, C peptide and glucose metrics | Baseline, 12 weeks
  Assessed by mixed meal testing.
Change in blood pressure | Baseline, 12 weeks
  Assessed by ambulatory blood pressure monitoring and home blood pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Kukla, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20557343